CLINICAL TRIAL: NCT05559723
Title: Effect of Electromagnetic Field Therapy on Sciatica and Postural Control in Lumbar Disc Prolapse Patients
Brief Title: Effect of Electromagnetic Field in Lumbar Disc Prolapse Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Lama Saad El-Din Mahmoud, Lecturer of physical therapy, Department of Neuromuscular disorders and its surgery, faculty of physical therapy, october 6 univerisity, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T. REC/012/004099
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Magnetic Field Therapy; Ultrasonic Therapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): electromagnetic field therapy
  Interventions: Device: electromagnetic field therapy; Other: selected physical therapy program; Device: Therapeutic ultrasound therapy; Device: Transcutaneous Electrical Nerve Stimulation
- control group (Experimental): the selected exercise program
  Interventions: Other: selected physical therapy program; Device: Therapeutic ultrasound therapy; Device: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Device: electromagnetic field therapy — Three times a week for four weeks, the study group got electromagnetic fields (EMFs) therapy and the selected physical therapy program. The EMFs therapy was applied using an electromagnetic field therapy device (Magner Plus Astar)
  . From the prone lying position the device will be adjusted around the lumbar area at a low frequency (50 Hz), with the intensity of 2.5 MT, field shape and applicator type rectangular csl60/csp60), and the application time will be10 minutes
  Arms: study group
Other: selected physical therapy program — in the form of
  1. Hot packs will be placed paravertebral on the lumbar region for 5 minutes from a prone lying position
  2. selected physical therapy exercises in form of Static exercise for back and abdominal muscles, stretching exercises for both lower limbs, 10 times each exercise
Device: Therapeutic ultrasound therapy — Therapeutic ultrasound therapy using ultrasound device Chattanooga, model 2760, serial number T11238, 120-240V, 50/60Hz, made in Mexico . That will be applied paravertebral on the lumbar region from the prone lying position, with pulsed mode, frequency 1 MHz, intensity 0.5 W/cm2 and will be applied by circular moving technique at a rate of 4 cm/s for 10 minutes.
Device: Transcutaneous Electrical Nerve Stimulation — Transcutaneous Electrical Nerve Stimulation (TENS): from the prone lying position, the electrodes will be placed on the course of pain detected by the patient, with an asymmetrical rectangular biphasic form, at a pulse repetition frequency of 100Hz and duty cycle of 250 microseconds; the intensity was set at a level that each patient could feel, for 15 minutes .

SUMMARY:
to investigate the effect of electromagnetic field therapy on sciatica and postural control in lumbar disc prolapse patients BACKGROUND: lumbar disc prolapse is a clinical condition resulting from compression of lumbar nerve roots resulting in decreased postural control and alleviating sciatic pain Pulsed electromagnetic field (PEMF) therapy is an easy, non-invasive, safe, and relatively new treatment method that is used with growing interest in physical and rehabilitation medicine. Historically, the benefits from magnetotherapy have been reported for patients with musculoskeletal and neurological disorders

DETAILED DESCRIPTION:
Thirty-four patients with lumbar disc prolapse The patients will randomly be divided into two equal groups; the control group which received the selected exercise program and the study group received the same exercise training program in addition to electromagnetic field therapy, three times per week for four weeks. The evaluation methods by Visual analogue scale for pain (VAS-P), ) multidirectional reach test, McGill pain Questionnaire, time up and go test and Oswestry Low Back Pain Disability Questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging from 30:45
2. sciatica due to lumbar disc prolapse mild to moderate disc prolapse according to magnetic resonance image (MRI).
3. Body mass index (18.5 to 29.9) Kg/m2.

Exclusion Criteria:

* The patients will be excluded if they have one of the followings:

  1. lumbar myelopathy.
  2. Patients with previous spinal surgery.
  3. Inflammatory diseases such as rheumatoid arthritis or ankylosing spondylitis
  4. Any other neurological or musculoskeletal disorders of the spine or upper extremity.
  5. Patient with cardiopulmonary disease or diabetes mellitus

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-11-25 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale | 4 weeks
  which assesses pain on a paper sheet scale with an increasing number from 0 (no pain) to 10 (the worst pain imaginable).
Multi-Directional Reach test | 4 weeks
  Multi-Directional Reach test (MDRT) is an assessment method used to evaluate the limits of stability of individuals in four directions "forward, backward, right and left".
  The normal Scores of the multi-directional reach test for individuals with age ranging from (20 to 39 cm) years are as follow: forward reach (28 cm); backward reach (17 to 18 cm); leftward reach (17 to 21 cm) and rightward reach (18 to 20 cm)
time up and go test | 4 weeks
  To determine fall risk and measure the progress of balance, sit to stand and walking.
  Simple screening test that is a sensitive and specific measure of probability for falls among older adults An older adult who takes ≥12 seconds to complete the TUG is at risk for falling
Oswestry Low Back Pain Disability Questionnaire | 4 weeks
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools For each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5. I

SECONDARY OUTCOMES:
The McGill Pain Questionnaire | four weeks
  The McGill Pain Questionnaire (MPQ) is a self-reporting measure of pain used for patients with a number of diagnoses. It assesses both quality and intensity of subjective pain. The MPQ is a multi-dimesional tool for pain assessment and it has three components, which are the sensory intensity, the cognitive evaluation of pain and the emotional impact of pain
  The MPQ is composed of 78 words, of which respondents choose those that best describe their experience of pain. Seven words are selected from the following categories: dimension 1 to 10 (pain descriptors), three words; dimensions 11 to 15 (affective components of pain), dimension 16 (evaluation of pain) one word, and dimension 17 to 20 (miscellaneous) one word. Scores are tabulated by summing values associated with each word; scores range from 0 (no pain) to 78 (severe pain). Qualitative differences in pain may be reflected in respondent's word choice

CONTACTS AND LOCATIONS:
Overall Officials: Lama Saad El-Din Mahmoud, PHD, Study Chair — October 6 University; KEROLOS AWAD HABIB SAEED, masters, Principal Investigator — October 6 University
Locations (1):
- Lama S Mahmoud, Al Jīzah, Select State, Egypt

IPD SHARING:
Plan to Share IPD: No